CLINICAL TRIAL: NCT02887157
Title: Analyzing Retinal Microanatomy in Retinopathy of Prematurity to Improve Care (BabySTEPS)
Brief Title: Analyzing Retinal Microanatomy in ROP
Acronym: BabySTEPS
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Eye Institute (NEI) (NIH); University of Pennsylvania (Other); Washington University School of Medicine (Other); University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00069721; R01EY025009-01A1 (NIH)
Record Dates: First submitted 2016-08-25; First posted 2016-09-02 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Retinopathy of Prematurity; Neurodevelopmental Disorders; Macular Edema
MeSH Terms: conditions — Retinopathy of Prematurity; Neurodevelopmental Disorders; Macular Edema | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum or plasma will be collected from scavenged blood (residual in the laboratory) collected as part of clinically indicated care. These samples will undergo neuroinflammatory biomarker testing to identify central nervous system cellular injury.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Specific Aim 1B: Specific Aim 1B (implement technical innovations to improve OCT imaging in non-sedated infants in the ICN: (1B) extend imaging to the vascular-avascular junction via a wide-field lens).
  Aim 1B only: 50 participants (25 healthy adult volunteers and 25 pediatric participants under going examination under anesthesia
  * Healthy adult volunteers will have SSOCT imaging of both eyes with the novel ultralight handpiece up to 10 times.
  * Pediatric participants undergoing examination under anesthesia will have SSOCT imaging of both eyes with the novel ultralight handpiece once during their EUA in the Duke Eye Center Operating Rooms (OR). These participants will be enrolled into the study at DUHS including the Duke Eye Center clinics and OR for testing the custom widefield lens.
  Interventions: Device: Swept Source OCT
- Specific Aim 2: Specific Aim 2 (distinguish elements of retinal microanatomy that predict maldevelopment of visual pathway and poor neurodevelopment that may impact vision in preterm infants) includes 68 very preterm infants undergoing the following during evaluation for ROP.
  1. Swept Source OCT imaging of both eyes with the novel ultralight handpiece before or after ROP examination, timed with each examination. The axial length of the eye may be measured after the ROP exam.
  2. Non-sedated research brain Magnetic Resonance Imaging will be obtained in 68 participants prior to discharge from the nursery whenever possible (as close to term age as possible). In the case of an early infant discharge to another hospital, every effort will be made to obtain brain MRI prior to transfer or an outpatient non-sedated brain MRI at near term age.
  3. Scavenged blood collection: Residual samples of serum/plasma in the laboratory will be collected for neuroinflammatory marker testing.
  Interventions: Device: Swept Source OCT; Other: Magnetic Resonance Imaging; Other: Scavenged blood collection
- Specific Aim 3: Specific Aim 3 (delineate which elements and regions (posterior) or (peripheral) of preterm infant OCT-derived retinal microanatomy best inform us about severity of disease and visual outcomes in infants with ROP will include the same 68 participants plus an additional 42 very preterm infants undergoing evaluation for ROP and visual function but who will not be in the neurodevelopmental study and thus will not have brain MRI, 2-year Bayley Scales testing or neuroinflammatory marker testing on scavenged blood. The Specific Aim 3 subjects will undergo the following:
  1. Swept Source OCT imaging of both eyes with the novel ultralight handpiece as described in Aim 2. The axial length of the eye may be measured after the ROP exam.
  2. After imaging with the original lens (ultralight handpiece) both eyes will be imaged with the widefield OCT lens. before or after the ROP exam.
  3. Ocular and systemic health data will be extracted from the study participant's medical record.
  Interventions: Device: Swept Source OCT

INTERVENTIONS:
Device: Swept Source OCT — The swept source optical coherence tomography device was developed at Duke University as the result of collaboration between the Departments of Ophthalmology and Biomedical Engineering. The SSOCT system has a 100kHz repetition rate, 1050nm-centered swept-source light source (Axsun Technologies). This swept-source system allows near real-time OCT imaging during movement while imaging and it provides better OCT imaging of the choroid. The SSOCT system is a non-contact device and therefore does not touch the eye.
  Other Names: SSOCT; Swept Source Optical Coherence Tomography
Other: Magnetic Resonance Imaging — Non-sedated research brain MRI: Magnetic resonance imaging (MRI) is a minimal risk procedure that uses a magnet and radio waves to make diagnostic medical images of the body. There have been no ill effects reported from exposure to the magnetism or radio waves used in this test. However, it is possible that harmful effects could be recognized in the future. A known risk is that the magnet could attract certain kinds of metal. Therefore, we will carefully ask about metal within the body. If there is any question about potentially hazardous metal within the body, MRI imaging will not be performed. We will also keep the examining room locked so that no one carrying metal objects can enter while the child is in the scanner.
  Other Names: MRI
  Groups: Specific Aim 2
Other: Scavenged blood collection — Serum/plasma (residual in the laboratory) collected as part of clinically indicated care will be shipped to the University of Florida for neuroinflammatory biomarker testing to identify central nervous system cellular injury.
  Groups: Specific Aim 2

SUMMARY:
Retinopathy of prematurity (ROP) is a disorder of development of the neural retina and its vasculature that may impact vision in vulnerable preterm neonates for a lifetime. This study utilizes new technology to determine visual and neurological development of very preterm infants in the intensive care nursery, during a period of rapid growth of the retina, optic nerve and brain. The long-term goal of this study is to help improve preterm infant health care via objective bedside imaging and analysis that characterizes early critical indicators of poor vision, neurological development and ROP, which will rapidly translate to better early intervention and improved future vision care.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is a disorder of development of the neural retina and its vasculature that may impact vision in vulnerable preterm neonates for a lifetime. Clinical care of infants with ROP decreases the likelihood of blindness, but abnormal vision is common, especially in those with disease severe enough to require treatment. Because it has not been possible to distinguish whether disease and/or maldevelopment that affects specific retinal cells and/or the central nervous system (CNS) cause the vision loss, especially when it is less severe, there has been no strategy to prevent subnormal acuity in the majority of infants treated for ROP.

The interval that a preterm infant at risk for ROP spends in an intensive care nursery (ICN) is a time of rapid retinal development. Clinicians and researchers do not know how local, CNS and systemic development and disease processes are reflected in the retinal microanatomy. Abnormalities in the retina during infancy are likely early predictors of later vision problems and developmental delay. From study of preterm retinal substructures, brain anatomy, connectivity and functional networks and neuroinflammatory biomarkers this study will elucidate the pathway by which local retinal anatomic changes impact and may predict later subnormal vision and CNS function. The results of this research will enable the investigator to: distinguish ocular from non-ocular contributions to vision loss; guide future treatment directed to modify retinal anomalies such as edema; and determine which microanatomic retinal biomarkers are best to monitor effects of ROP, and effects of systemic therapies on the eye and brain. In contrast to indirect ophthalmoscopy or photography, novel non-contact ocular imaging at the bedside would enable direct telemedicine screening for ROP and for neural development in multiple nurseries.

The long-term goal is to help improve preterm infant health care via objective bedside imaging and analysis that characterizes early critical indicators of poor vision, neurological development and ROP. This will rapidly translate to early intervention and improved future vision care. Specific goals of this research are threefold: to implement technological innovations to improve optical coherence tomography (OCT) imaging in non-sedated infants in the ICN; to distinguish elements of retinal microanatomy which predict maldevelopment of visual pathway and poor neurodevelopment that may impact vision in preterm infants; and to delineate which elements and regions (posterior and peripheral) of preterm infant OCT-derived retinal microanatomy best inform us about severity of disease and visual outcomes in infants with ROP.

In addition to providing a breakthrough method for bedside analysis of the very preterm (VPT) infant posterior and peripheral retina, this study will provide the pediatric ophthalmologic and telemedicine community with methods to distinguish microanatomic markers that predict infants at risk for abnormal vision, visual pathway injury, poor functional development and progression of ROP (and combinations thereof). These biomarkers will be useful for determining ophthalmic and CNS therapeutic interventions and monitoring their impact on the visual pathway and will thus likely cross over with relevance to other infant eye and brain disease.

ELIGIBILITY:
Inclusion Criteria:

* Health care provider, knowledgeable of protocol, agrees that study personnel could contact the Parent/Legal Guardian
* Parent/Legal Guardian is able and willing to consent to study participation for the infant with likelihood of follow up at standard of care visits at approximately 1-month, 4-months, 9-months and 2 years corrected age
* Infant/child undergoing clinically indicated examination under anesthesia (for the testing of the custom widefield OCT lens) that may or may not have eye pathology. (Only for Aim 1)
* Infant meets the American Association of Pediatrics eligibility of ROP screening (Infants with a birth weight of ≤1500 g or gestational age of 30 weeks), and is age ≤ 34 6/7 weeks postmenstrual age at first visit
* Adults (over the age of 18 years) that may or may not have eye pathology (Only for Aim *Participants in Aim 3 will not have a brain MRI, collection of scavenged blood for neuroinflammatory markers, or the neurodevelopmental 2-year visit.

Exclusion Criteria:

* Participant or Parent/Legal Guardian (of infant/child) unwilling or unable to provide consent
* Adult participant or infant/child has a health or eye condition that preclude eye examination or retinal imaging (e.g. corneal opacity such as with Peters anomaly or cataract)
* Infant has a health condition, other than prematurity, that has a profound impact on brain development (e.g. anencephaly). Note that infants with brain hemorrhages and sequelae would be eligible.

Min Age: 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will have approximately 160 participants recruited and consented into the study at Duke University Health System. Of the 160 participants, 135 will be pediatric participants (of which 110 will be infants in the ICN) and 25 will be healthy adult volunteers. Infants in the ICN must meet the American Association of Pediatrics eligibility of ROP screening (Infants with a birth weight of ≤1500 g or gestational age of 30 weeks), and is age ≤ 34 6/7 weeks postmenstrual age at first visit.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Initiate ICN research imaging with the novel ultralight hand piece and high speed SSOCT (Aim 1A) | 4 years
  Start-up of research imaging in the intensive care nursery using the new ultralight hand piece and swept source OCT
Number of infants with reproducible imaging of the peripheral vascular-avascular junction (Aim 1B) | 4 years
  Analysis of reproducibility of imaging of the peripheral vascular-avascular junction in infants
Number of microns of retinal thickness and distance from foveal to ellipsoid zone band as seen on retinal vascular imaging using infant specific automated image processing | 3 months
  Develop infant-specific automated image processing/analyses for retinal vascular imaging
Number of microns of retinal thickness and distance from foveal to ellipsoid zone band as seen from multi-layer segmentation using infant specific automated image processing (1C) | 3 months
  Develop infant-specific automated image processing/analyses or multi-layer segmentation
Retinal microanatomy grading from Swept Source Optical Coherence Tomography (SSOCT) | 4 years
  Grading and measurement of retinal microanatomy from SSOCT images
Brain MRI grading | 3 years
  Grading and analysis of brain MRI scans collected at approximately term-equivalent age
Visual acuity scores | 3 years
  Analyses of data from Teller Visual acuity testing at 9 months
Neurodevelopmental scores | 3 years
  Analysis of Bayley Scales-III Neurodevelopmental testing at age 2 years
Peripheral retinal microanatomy grading | 4 years
  Analyses of peripheral retinal microanatomy at the vascular-avascular junction as recorded via SSOCT
ROP severity grade of retinal microanatomy by OCT | 4 years
  Severity of ROP as determined by analysis of posterior and peripheral retinal microanatomy
Maximum ROP stage as determined during clinical evaluation | 4 years
  Analysis of maximum ROP stage per eye as determined during clinical evaluation

SECONDARY OUTCOMES:
Neuroinflammatory marker scores | 2 years
  Analysis of left over blood samples to determine presence and severity of neuroinflammation
Presence of non-ROP ocular conditions | 4 years
  Analysis of clinical data for strabismus,, amblyopia, refractive error, nystagmus
ROP specifics from clinical examination | 4 years
  ROP specifics including zone, plus or preplus disease, stage per clock hour, vitreous hemorrhage from clinical examination
ROP specifics from OCT imaging | 4 years
  ROP specifics including zone, plus or preplus disease, stage per clock hour, vitreous hemorrhage from OCT imaging
Clinician's decision to treat | 4 years
  Analysis of the clinician's decision to treat

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Toth, MD, Principal Investigator — Duke Health
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Washington University, St Louis, Missouri
  - Duke University Eye Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Chen X, Mangalesh S, Tran-Viet D, Freedman SF, Vajzovic L, Toth CA. Fluorescein Angiographic Characteristics of Macular Edema During Infancy. JAMA Ophthalmol. 2018 May 1;136(5):538-542. doi: 10.1001/jamaophthalmol.2018.0467. PMID 29621379
- [Background] Lee J, El-Dairi MA, Tran-Viet D, Mangalesh S, Dandridge A, Jiramongkolchai K, Viehland C, Toth CA. LONGITUDINAL CHANGES IN THE OPTIC NERVE HEAD AND RETINA OVER TIME IN VERY YOUNG CHILDREN WITH FAMILIAL EXUDATIVE VITREORETINOPATHY. Retina. 2019 Jan;39(1):98-110. doi: 10.1097/IAE.0000000000001930. PMID 29190238
- [Background] Tran-Viet D, Wong BM, Mangalesh S, Maldonado R, Cotten CM, Toth CA. HANDHELD SPECTRAL DOMAIN OPTICAL COHERENCE TOMOGRAPHY IMAGING THROUGH THE UNDILATED PUPIL IN INFANTS BORN PRETERM OR WITH HYPOXIC INJURY OR HYDROCEPHALUS. Retina. 2018 Aug;38(8):1588-1594. doi: 10.1097/IAE.0000000000001735. PMID 28570486
- [Background] Rothman AL, Mangalesh S, Chen X, Toth CA. Optical coherence tomography of the preterm eye: from retinopathy of prematurity to brain development. Eye Brain. 2016 May 27;8:123-133. doi: 10.2147/EB.S97660. eCollection 2016. PMID 28539807
- [Background] Mangalesh S, Chen X, Tran-Viet D, Viehland C, Freedman SF, Toth CA. ASSESSMENT OF THE RETINAL STRUCTURE IN CHILDREN WITH INCONTINENTIA PIGMENTI. Retina. 2017 Aug;37(8):1568-1574. doi: 10.1097/IAE.0000000000001395. PMID 28085775
- [Background] Ong SS, Mruthyunjaya P, Stinnett S, Vajzovic L, Toth CA. Macular Features on Spectral-Domain Optical Coherence Tomography Imaging Associated With Visual Acuity in Coats' Disease. Invest Ophthalmol Vis Sci. 2018 Jun 1;59(7):3161-3174. doi: 10.1167/iovs.18-24109. PMID 30025132
- [Background] Finn AP, Chen X, Viehland C, Izatt JA, Toth CA, Vajzovic L. COMBINED INTERNAL LIMITING MEMBRANE FLAP AND AUTOLOGOUS PLASMA CONCENTRATE TO CLOSE A LARGE TRAUMATIC MACULAR HOLE IN A PEDIATRIC PATIENT. Retin Cases Brief Rep. 2021 Mar 1;15(2):107-109. doi: 10.1097/ICB.0000000000000762. PMID 29979253
- [Background] Hsu ST, Chen X, House RJ, Kelly MP, Toth CA, Vajzovic L. Visualizing Macular Microvasculature Anomalies in 2 Infants With Treated Retinopathy of Prematurity. JAMA Ophthalmol. 2018 Dec 1;136(12):1422-1424. doi: 10.1001/jamaophthalmol.2018.3926. No abstract available. PMID 30326081
- [Background] Ong SS, Cummings TJ, Vajzovic L, Mruthyunjaya P, Toth CA. Comparison of Optical Coherence Tomography With Fundus Photographs, Fluorescein Angiography, and Histopathologic Analysis in Assessing Coats Disease. JAMA Ophthalmol. 2019 Feb 1;137(2):176-183. doi: 10.1001/jamaophthalmol.2018.5654. PMID 30476946
- [Background] Hsu ST, Chen X, Ngo HT, House RJ, Kelly MP, Enyedi LB, Materin MA, El-Dairi MA, Freedman SF, Toth CA, Vajzovic L. Imaging Infant Retinal Vasculature with OCT Angiography. Ophthalmol Retina. 2019 Jan;3(1):95-96. doi: 10.1016/j.oret.2018.06.017. Epub 2018 Jul 26. No abstract available. PMID 30935662
- [Background] Mangalesh S, Bleicher ID, Chen X, Viehland C, LaRocca F, Izatt JA, Freedman SF, Hartnett ME, Toth CA. Three-dimensional pattern of extraretinal neovascular development in retinopathy of prematurity. Graefes Arch Clin Exp Ophthalmol. 2019 Apr;257(4):677-688. doi: 10.1007/s00417-019-04274-6. Epub 2019 Feb 21. PMID 30790072
- [Background] Smith LEH, Hellstrom A, Stahl A, Fielder A, Chambers W, Moseley J, Toth C, Wallace D, Darlow BA, Aranda JV, Hallberg B, Davis JM; Retinopathy of Prematurity Workgroup of the International Neonatal Consortium. Development of a Retinopathy of Prematurity Activity Scale and Clinical Outcome Measures for Use in Clinical Trials. JAMA Ophthalmol. 2019 Mar 1;137(3):305-311. doi: 10.1001/jamaophthalmol.2018.5984. PMID 30543348
- [Background] Hsu ST, Ngo HT, Stinnett SS, Cheung NL, House RJ, Kelly MP, Chen X, Enyedi LB, Prakalapakorn SG, Materin MA, El-Dairi MA, Jaffe GJ, Freedman SF, Toth CA, Vajzovic L. Assessment of Macular Microvasculature in Healthy Eyes of Infants and Children Using OCT Angiography. Ophthalmology. 2019 Dec;126(12):1703-1711. doi: 10.1016/j.ophtha.2019.06.028. Epub 2019 Jul 15. PMID 31548134
- [Background] Mangalesh S, Tran-Viet D, Pizoli C, Tai V, El-Dairi MA, Chen X, Viehland C, Edwards L, Finkle J, Freedman SF, Toth CA. Subclinical Retinal versus Brain Findings in Infants with Hypoxic Ischemic Encephalopathy. Graefes Arch Clin Exp Ophthalmol. 2020 Sep;258(9):2039-2049. doi: 10.1007/s00417-020-04738-0. Epub 2020 May 29. PMID 32472201
- [Background] Cai CX, Go M, Kelly MP, Holgado S, Toth CA. OCULAR MANIFESTATIONS OF PORETTI-BOLTSHAUSER SYNDROME: FINDINGS FROM MULTIMODAL IMAGING AND ELECTROPHYSIOLOGY. Retin Cases Brief Rep. 2022 May 1;16(3):270-274. doi: 10.1097/ICB.0000000000000991. Epub 2020 Mar 17. PMID 32195884
- [Result] Viehland C, Chen X, Tran-Viet D, Jackson-Atogi M, Ortiz P, Waterman G, Vajzovic L, Toth CA, Izatt JA. Ergonomic handheld OCT angiography probe optimized for pediatric and supine imaging. Biomed Opt Express. 2019 Apr 29;10(5):2623-2638. doi: 10.1364/BOE.10.002623. eCollection 2019 May 1. PMID 31143506
- [Result] Chen X, Viehland C, Tran-Viet D, Prakalapakorn SG, Freedman SF, Izatt JA, Toth CA. Capturing Macular Vascular Development in an Infant With Retinopathy of Prematurity. JAMA Ophthalmol. 2019 Sep 1;137(9):1083-1086. doi: 10.1001/jamaophthalmol.2019.2165. No abstract available. PMID 31246250
- [Result] Chen X, Mangalesh S, Dandridge A, Tran-Viet D, Wallace DK, Freedman SF, Toth CA. Spectral-Domain OCT Findings of Retinal Vascular-Avascular Junction in Infants with Retinopathy of Prematurity. Ophthalmol Retina. 2018 Sep;2(9):963-971. doi: 10.1016/j.oret.2018.02.001. Epub 2018 Mar 21. PMID 30506013
- [Result] Chen X, Prakalapakorn SG, Freedman SF, Vajzovic L, Toth CA. Differentiating Retinal Detachment and Retinoschisis Using Handheld Optical Coherence Tomography in Stage 4 Retinopathy of Prematurity. JAMA Ophthalmol. 2020 Jan 1;138(1):81-85. doi: 10.1001/jamaophthalmol.2019.4796. PMID 31774474
- [Result] Wang KL, Chen X, Stinnett S, Tai V, Winter KP, Tran-Viet D, Toth CA. Understanding the variability of handheld spectral-domain optical coherence tomography measurements in supine infants. PLoS One. 2019 Dec 11;14(12):e0225960. doi: 10.1371/journal.pone.0225960. eCollection 2019. PMID 31825990
- [Result] Seely KR, Wang KL, Tai V, Prakalapakorn SG, Chiu SJ, Viehland C, Grace S, Izatt JA, Freedman SF, Toth CA. Auto-Processed Retinal Vessel Shadow View Images From Bedside Optical Coherence Tomography to Evaluate Plus Disease in Retinopathy of Prematurity. Transl Vis Sci Technol. 2020 Aug 7;9(9):16. doi: 10.1167/tvst.9.9.16. eCollection 2020 Aug. PMID 32879772
- [Result] Mangalesh S, McGeehan B, Tai V, Chen X, Tran-Viet D, Vajzovic L, Viehland C, Izatt JA, Cotten CM, Freedman SF, Maguire MG, Toth CA; Study of Eye Imaging in Preterm Infants Group. Macular OCT Characteristics at 36 Weeks' Postmenstrual Age in Infants Examined for Retinopathy of Prematurity. Ophthalmol Retina. 2021 Jun;5(6):580-592. doi: 10.1016/j.oret.2020.09.004. Epub 2020 Sep 11. PMID 32927150
- [Result] Shen LL, Mangalesh S, McGeehan B, Tai V, Sarin N, El-Dairi MA, Freedman SF, Maguire MG, Toth CA; BabySTEPS Group. Birth Weight Is a Significant Predictor of Retinal Nerve Fiber Layer Thickness at 36 Weeks Postmenstrual Age in Preterm Infants. Am J Ophthalmol. 2021 Feb;222:41-53. doi: 10.1016/j.ajo.2020.08.043. Epub 2020 Sep 4. PMID 32891695
- [Result] Chen X, Tai V, McGeehan B, Ying GS, Viehland C, Imperio R, Winter KP, Raynor W, Tran-Viet D, Mangalesh S, Maguire MG, Toth CA; BabySTEPS Group. Repeatability and Reproducibility of Axial and Lateral Measurements on Handheld Optical Coherence Tomography Systems Compared with Tabletop System. Transl Vis Sci Technol. 2020 Oct 21;9(11):25. doi: 10.1167/tvst.9.11.25. eCollection 2020 Oct. PMID 33150050
- [Result] Mangalesh S, Wong BM, Chen X, Tran-Viet D, Stinnett SS, Sarin N, Winter KP, Vajzovic L, Freedman SF, Toth CA. Morphological characteristics of early- versus late-onset macular edema in preterm infants. J AAPOS. 2020 Oct;24(5):303-306. doi: 10.1016/j.jaapos.2020.06.006. Epub 2020 Sep 15. PMID 32942022
- [Result] Chen X, Imperio R, Seely KR, Viehland C, Izatt JA, Prakalapakorn SG, Freedman SF, Toth CA. Slow progressive perifoveal vascular formation in an infant with aggressive posterior retinopathy of prematurity. J AAPOS. 2020 Oct;24(5):323-326. doi: 10.1016/j.jaapos.2020.07.007. Epub 2020 Oct 9. PMID 33045380
- [Result] O'Sullivan ML, Ying GS, Mangalesh S, Tai V, Divecha HR, Winter KP, Toth CA, Chen X; BabySTEPS Group. Foveal Differentiation and Inner Retinal Displacement Are Arrested in Extremely Premature Infants. Invest Ophthalmol Vis Sci. 2021 Feb 1;62(2):25. doi: 10.1167/iovs.62.2.25. PMID 33599735
- [Result] Prakalapakorn SG, Sarin N, Sarin N, McGeehan B, Tran-Viet D, Tai V, Ying GS, Toth CA, Freedman SF. Evaluating the association of clinical factors and optical coherence tomography retinal imaging with axial length and axial length growth among preterm infants. Graefes Arch Clin Exp Ophthalmol. 2021 Sep;259(9):2661-2669. doi: 10.1007/s00417-021-05158-4. Epub 2021 Mar 29. PMID 33779799
- [Result] Mangalesh S, Sarin N, McGeehan B, Prakalapakorn SG, Tran-Viet D, Cotten CM, Freedman SF, Maguire MG, Toth CA; BabySTEPS Group. Preterm Infant Stress During Handheld Optical Coherence Tomography vs Binocular Indirect Ophthalmoscopy Examination for Retinopathy of Prematurity. JAMA Ophthalmol. 2021 May 1;139(5):567-574. doi: 10.1001/jamaophthalmol.2021.0377. PMID 33792625
- [Result] Patel PR, Imperio R, Viehland C, Tran-Viet D, Chiu SJ, Tai V, Izatt JA, Toth CA, Chen X; BabySTEPS Group. Depth-Resolved Visualization of Perifoveal Retinal Vasculature in Preterm Infants Using Handheld Optical Coherence Tomography Angiography. Transl Vis Sci Technol. 2021 Aug 2;10(9):10. doi: 10.1167/tvst.10.9.10. PMID 34357383
- [Result] Shen LL, Mangalesh S, Michalak SM, McGeehan B, Sarin N, Finkle J, Winter KP, Tran-Viet D, Benner EJ, Vajzovic L, Freedman SF, Younge N, Cotten CM, El-Dairi M, Ying GS, Toth C. Associations between systemic health and retinal nerve fibre layer thickness in preterm infants at 36 weeks postmenstrual age. Br J Ophthalmol. 2023 Feb;107(2):242-247. doi: 10.1136/bjophthalmol-2021-319254. Epub 2021 Aug 13. PMID 34389548
- [Result] Mangalesh S, Seely KR, Tran-Viet D, Tai V, Chen X, Prakalapakorn SG, Freedman SF, Toth CA; BabySTEPS Group. Integrated Visualization Highlighting Retinal Changes in Retinopathy of Prematurity From 3-Dimensional Optical Coherence Tomography Data. JAMA Ophthalmol. 2022 Jul 1;140(7):725-729. doi: 10.1001/jamaophthalmol.2022.1344. PMID 35616956
- [Result] Seely KR, Mangalesh S, Shen LL, McGeehan B, Ying GS, Sarin N, Vajzovic L, Prakalapakorn SG, Freedman SF, Toth CA; BabySTEPS Group. Association Between Retinal Microanatomy in Preterm Infants and 9-Month Visual Acuity. JAMA Ophthalmol. 2022 Jul 1;140(7):699-706. doi: 10.1001/jamaophthalmol.2022.1643. PMID 35653144
- [Result] Seely KR, Weinert MC, Hong GJ, Wang W, Grace S, Freedman SF, Toth CA, Prakalapakorn SG. Semi-automated vessel analysis of en face posterior pole vessel maps generated from optical coherence tomography for diagnosis of plus or pre-plus disease. J AAPOS. 2022 Aug;26(4):199-202. doi: 10.1016/j.jaapos.2022.03.008. Epub 2022 Jun 3. PMID 35667618
- [Result] Shen LL, Mangalesh S, McGeehan B, Seely KR, Tai V, Sarin N, Finkle J, Winter KP, Tran-Viet D, Freedman SF, El-Dairi MA, Ying GS, Toth CA. Biphasic change in retinal nerve fibre layer thickness from 30 to 60 weeks postmenstrual age in preterm infants. Br J Ophthalmol. 2023 Nov;107(11):1680-1686. doi: 10.1136/bjo-2022-321621. Epub 2022 Sep 16. PMID 36113954
- [Result] Michalak SM, Mangalesh S, Shen LL, McGeehan B, Winter KP, Sarin N, Finkle J, Cotten M, Ying GS, Toth CA, Vajzovic L. Systemic Factors Associated with a Thinner Choroid in Preterm Infants. Ophthalmol Sci. 2021 Jun 7;1(2):100032. doi: 10.1016/j.xops.2021.100032. eCollection 2021 Jun. PMID 36249299